CLINICAL TRIAL: NCT06534671
Title: Diltiazem in Jervell and Lange-Nielsen Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Prince Joseph Kannankeril, Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 240535
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Jervell and Lange Nielsen Syndrome
Keywords: Long QT syndrome
MeSH Terms: conditions — Jervell-Lange Nielsen Syndrome; Long QT Syndrome | interventions — Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diltiazem (Experimental): IV diltiazem (0.25 mg/kg) will be given over 2 minutes. A second IV dose (0.35 mg/kg) may be given at 10 minutes.
  Interventions: Drug: diltiazem

INTERVENTIONS:
Drug: diltiazem — IV diltiazem (0.25 mg/kg) will be given over 2 minutes, with ECG and blood pressure measurements at baseline, 2, 5, 7, 10, 15 and 20 minutes. If at 10 minutes there is no QT shortening, and blood pressure is stable, an additional dose (0.35 mg/kg) will be given with ECG and blood pressure measurements at 17, 20, 22, 25, 30 and 35 minutes.

SUMMARY:
This study will test the effect of diltiazem, a calcium channel blocking drug, on the QT interval in patients with Jervell and Lange-Nielsen syndrome. This will be a single IV dose and acute effects (within minutes) will be observed.

DETAILED DESCRIPTION:
Subjects will be recruited by study personnel and will be scheduled for a single outpatient visit. If an implanted cardiac device (pacemaker or ICD) is in place, it will be interrogated to ensure no recent rhythm abnormalities. Just prior to administering diltiazem, an ECG and BP will be obtained. If baseline SBP is < 100 mm Hg or DBP < 60 mm Hg, the study will be terminated. A single dose of I.V. diltiazem (0.25 mg/kg over 2 minutes) will be administered with 12-lead ECG and BP obtained at 2, 5, 7, 10, 15 and 20 minutes. If at 10 minutes there has been no QT shortening, and the SBP is stable (<20% drop from baseline and > 100 mm Hg) a repeat dose (0.35 mg/kg) will be given at 15 minutes, with 12-lead ECG and BP obtained at 17, 20, 22, 25, 30 and 35 minutes. After 20 minutes (single dose) or 35 minutes (2 doses), the test will end and the subject will remain on continuous telemetry for 2 hours. Prior to discharge the IV will be removed. The primary analysis will be a repeated measures (paired) comparison of the QTc at baseline and following diltiazem.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Genetically confirmed diagnosis of Jervell and Lange-Nielsen syndrome
* Able to provide written informed consent

Exclusion Criteria:

* Known hypersensitivity to diltiazem
* Pregnancy
* Congestive heart failure, angina, preexcitation, or chronic obstructive pulmonary disease
* Sick sinus syndrome or atrioventricular block in the absence of a pacemaker/defibrillator
* Any clinically significant ongoing medical or surgical condition that might jeopardize the subject's safety or interfere with the conduct of the study in the judgement of the investigator
* Baseline systolic blood pressure less than 100 Hg or diastolic blood pressure less than 60 Hg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prince J Kannankeril, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual-level QT results will be published. Data obtained through this study may be provided to qualified researchers with no PHI included.
Time Frame: Data requests can be submitted immediately after article publication and the data will be made accessible for up to 36 months.
Access Criteria: Access may be requested by qualified researchers and will be provided following review and approval of a research proposal and execution of a Data Use Agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diltiazem
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diltiazem
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] — Years
  years | 29 [29 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: QT Interval
Description: QT interval (on 12-lead ECG) in ms
Time Frame: Baseline
Measure: Number; unit: ms
Arm/Group | Diltiazem
Number analyzed (Participants) | 1
ms | 623

2. Primary Outcome: QT Interval
Description: QT interval (on 12-lead ECG) in ms
Time Frame: 5 minutes
Measure: Number; unit: ms
Arm/Group | Diltiazem
Number analyzed (Participants) | 1
ms | 570

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Diltiazem
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT06534671/Prot_002.pdf
  • Informed Consent Form (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT06534671/ICF_000.pdf